CLINICAL TRIAL: NCT00940537
Title: MRS Validation Study of Hepatic Triglyceride Content in Non-alcoholic Fatty Liver Disease (NAFLD)Subjects Pre- and Post-Prandial
Brief Title: Magnetic Resonance Spectroscopy (MRS) Validation Study in Individuals With Nonalcoholic Fatty Liver Disease (NAFLD)
Acronym: NAFLD
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 06-0229
Record Dates: First submitted 2009-07-14; First posted 2009-07-16 (Estimated); Results first posted 2010-05-13 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Liver Diseases
Keywords: Obese; MRS; hepatic triglyceride content; MR spectroscopy
MeSH Terms: conditions — Liver Diseases; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NAFLD: Non-diabetic, obese with diagnosed NAFLD (HTGC greater or equal to 5.5%)
- Non-NAFLD: Non-diabetic, obese with no previous diagnosis of NAFLD

SUMMARY:
The purpose of this study is to see how effective the investigators' optimized magnetic resonance spectroscopy (MRS) sequence in quantifying hepatic triglyceride content (HTGC) to enhance MRS as a diagnostic tool in non-alcohol fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
One way to gauge MRS as an effective diagnostic tool is by looking at the reproducibility of the liver fat measurements on subjects by calculating the coefficient of variation (CV). This study assesses the modified MRS sequence, using both breath holds and free breathing. The HTGC levels are measured twice in the same individuals on two independent events separated by 10 minutes. Subjects are then given a high fat, high carbohydrate meal of Pizza Hut pizza, Pepsi, and Oreo cookies. Two hours after eating the meal, the subjects return to the scanner and repeat all MRS scans.

ELIGIBILITY:
Inclusion Criteria:

* Obese

Exclusion Criteria:

* Diabetes
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: St. Louis community
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, M.D., Principal Investigator — Washinton University in St. Louis
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through the Center for Human Nutrition (CHN) beginning in July, 2009. Many had previously been enrolled in other CHN studies. The final subject was tested in December, 2009.
Pre-assignment Details: All enrolled subjects completed the study.
Groups:
- NAFLD: Non-diabetic, obese with diagnosed NAFLD (hepatic triglyceride content (HTGC) greater or equal to 5.5%)
Period: Overall Study
Arm/Group | NAFLD | Non-NAFLD
Started | 5 | 9
Completed | 5 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NAFLD | Non-NAFLD | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 8 | 13
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (13) | 46 (12) | 45 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: The Reproducibility of the Hepatic Triglyceride Content Measurement by MRS.
Description: We compared three 1H-Magnetic Resonance Spectroscopy sequences: A Standard Siemens sequence, and an optimized sequence with either breath-holds or free-breathing. Repeat scans were done with the subject briefly removed from and returned to the scanner between scans. The results given are coefficients of variation of the triglyceride signal divided by the water signal.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: coefficient of variation
Arm/Group | NAFLD | Non-NAFLD
Number analyzed (Participants) | 5 | 9
coefficient of variation
  Siemens sequence | 13.0 (9.6) | 23.5 (1.1)
  Optimized sequence | 4.4 (3.9) | 9.7 (0.1)

2. Secondary Outcome: The Hepatic Triglyceride Content Pre- and Post-prandial.
Description: We compared the intrahepatic triglyceride content in subjects after a 12 hour fast and 2 hours after eating a high fat, high carbohydrate meal. The measure reported here is for the pre and post prandial results given as the ratio of triglyceride signal to water signal. After showing its reliability, we chose to use the results from the optimized breath-hold sequence.
Time Frame: after a 12 hour fast and 2 hours post-prandial
Measure: Mean (Standard Error); unit: ratio
Arm/Group | NAFLD | Non-NAFLD
Number analyzed (Participants) | 5 | 9
ratio
  fasting | 30 (12) | 8 (7)
  post-prandial | 27 (9) | 8 (7)
Statistical Analysis 1: Comparison: NAFLD vs Non-NAFLD; As there was no a priori reason for the level of IHTG to impact this measurement we compared the pre and post-prandial results for all subjects whose data were of sufficient quality (N=12). These results are comparing the two categories of fasting and post-prandial. Null hypothesis was that there would be no difference in IHTG before and after a high fat, high carbohydrate meal; Test type: Superiority or Other; p = .097, t-test, 2 sided — a priori threshhold for significance was set at p<0.05; this was a paired t-test

3. Secondary Outcome: T2 (Spin-spin Relaxation Time) Ratios of Triglyceride/Water
Description: T2 (spin-spin relaxation time) ratios of triglyceride/water using optimized PRESS sequences
Time Frame: baseline cross-sectional measurements
Population: This analysis was per protocol.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- All Subjects: all subjects studied. This includes both lean and obese subjects with a range of intrahepatic triglyceride.
Arm/Group | All Subjects
Number analyzed (Participants) | 14
ratio
  Low IHTG | 0.9 (0.1)
  Medium IHTG | 1.1 (0.1)
  High IHTG | 1.1 (0.1)
Statistical Analysis 1: Comparison: All Subjects; null hypothesis was that the T2 ratio would not depend on level of intrahepatic triglyceride (IHTG) and would be equal for the low and medium IHTG categories; Test type: Superiority or Other; p = 0.006, t-test, 2 sided — This p-value compares the low IHTG (<5%) subjects to those with medium levels of IHTG (5 - 10%). The a priori threshold for statistical significance was p<0.05
Statistical Analysis 2: Comparison: All Subjects; null hypothesis was that the T2 ratio would not depend on level of intra-hepatic triglyceride (IHTG) and would be equal for the low (<5%) and high (>10%) IHTG categories; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — The a priori threshold for statistical significance was p<0.05
Statistical Analysis 3: Comparison: All Subjects; The null hypothesis was that there would be no difference in T2 relaxation ratios for varying levels of intra-hepatic triglyceride (IHTG). Thus the medium (5 - 10%) and high (<10%) IHTG groups would not be statistically different with regard to average T2 ratio; Test type: Superiority or Other; p = .93, t-test, 2 sided — The a priori threshold for statistical significance was set at p<0.05

ADVERSE EVENTS:
Arm/Group | NAFLD | Non-NAFLD
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 0/5 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No